CLINICAL TRIAL: NCT03669094
Title: Randomized, Multicenter, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Effectiveness of the Strain Lactobacillus Salivarius V4II-90 in the Reduction of Group B Streptococcus Colonization in Pregnant Women
Brief Title: Effect of a New Probiotic Strain in the Reduction of Group B Streptococcus Colonization in Pregnant Women
Acronym: PROBIGEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProbiSearch SL (Industry)
Collaborators: Casen Recordati S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STB/17.02
Record Dates: First submitted 2018-08-30; First posted 2018-09-13 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Gestational Mother; Streptococcus Agalactiae Infection
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Intervention Model Description: This is an interventional randomized, multicenter, double-blind, placebo-controlled, parallel-group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L. salivarius V4II-90 (Active Comparator): Lactobacillus salivarius V4II-90; approximately 1*10E9 colony forming unit (CFU) of L. salivarius V4II-90 in 1 oral capsule per day for 12 weeks.
  Interventions: Dietary Supplement: Lactobacillus salivarius V4II-90
- Control group (Placebo Comparator): Placebo supplement in 1 oral capsule per day for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus salivarius V4II-90 — 7 months intervention study: with a screening period of 12 weeks after which participants GBS+ women will be randomized and start the orally intake of 1 capsule per day of the Lactobacillus salivarius V4II-90 (1*10E9 CFU) probiotic supplement over a 12 weeks period. A visit will then be completed one month after delivery.
  Arms: L. salivarius V4II-90
Dietary Supplement: Placebo — 7 months intervention study: with a screening period of 12 weeks after which participants GBS+ women will be randomized and start the orally intake of 1 capsule per day of the placebo supplement over a 12 weeks period. A visit will then be completed one month after delivery.
  Arms: Control group

SUMMARY:
An interventional, randomized, multicenter, double-blind, placebo-controlled, parallel-group study will be conducted to evaluate the effectiveness of the strain Lactobacillus salivarius V4II-90 in the reduction of Group B Streptococcus (GBS) colonization in pregnant women who are GBS carriers. Forty GBS-positive participants in their first trimester of pregnancy will be randomly assigned to one of the two study groups: The experimental group with 3 months probiotic consumption; and the control group with 3 months placebo consumption. The efficacy of the probiotic strain to reduce the incidence of Group B Streptococcus will be assessed by the percentage of participants with a vaginal and/or rectal detection of Group B Streptococcus at the end of the study, by bilateral comparison of the treatment group with the control group at the same time period. The estimated duration of the study will be 30 weeks, which includes a 3-month product administration. The intervention will start at week 23 ± 4 days of pregnancy and end at week 35 ± 4 days. Then, a visit will be completed one month after delivery.

DETAILED DESCRIPTION:
All pregnant women reporting to the clinic in their first trimester of pregnancy (week 11 ± 2 weeks of pregnancy) will be asked to participate in this study. Participation will be voluntary and written informed consent will be obtained from each participant. The study visits will take place in the hospital.

At Visit 1, the inclusion and exclusion criteria will be verified. After signing the informed consent, a physical examination will be performed in addition to a vaginal-rectal smear to detect if they are GBS-positive. Information on the demographic profile and medical history will be collected. The investigator will explain to the participant that she cannot use any probiotic during the course of the study.

At Visit 2, within 21-23 weeks ± 4 days of gestation, the inclusion and exclusion criteria will be reviewed. When a positive result of the microbiological analysis of the vaginal-rectal exudate are obtained, the pregnant GBS+ women will be invited to continue in the study. The randomized participant will intake one capsule of probiotic or placebo every day for the next 12 weeks. The participant will be given a diary and instructions to record the product intake. Adverse events occurring from the time of study inclusion will be recorded. Adverse Events occurring from the time of study inclusion will be recorded.

At the third visit (Visit 3, 35 weeks ± 4 days of gestation), all participants continuing in the study will undergo a general physical examination. A sample of vaginal and rectal exudate will be collected from the participants who end the treatment period. Adverse Events occurring during the period between Visit 2 and Visit 3 will be recorded. The participants must deliver the remaining product and the completed diary.

During Visit 4 (1 month after delivery), all participants will have a general physical examination. Adverse Events occurring since Visit 3 will be recorded. Data will be collected on the delivery and occurrence of early- or late-onset GBS sepsis in the newborn during the first month of life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women, adults (≥ 18 years and under 45 years).
* Before/during week 13 of gestation.
* Signing of informed consent.

Exclusion Criteria:

* Multiple pregnancy.
* Fetal complications.
* History of premature delivery/miscarriage in the second trimester.
* Significant maternal medical complications.
* HIV-positive.
* Women who are immunocompromised (for example, patients with cancer and transplant who are taking certain immunosuppressive drugs, patients with hereditary diseases that affect or could affect the immune system).
* History of significant gastrointestinal disease (e.g., prior gastrointestinal resection, current diarrhea, inflammatory bowel disease).
* Heart failure and cardiac medical history (e.g. artificial heart valve, medical history of infective endocarditis, rheumatic fever or cardiac malformation).
* Use of other probiotics during the current pregnancy.
* Uncertainty of the investigator regarding the willingness or capacity of the participant to comply with the requirements of the protocol.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 40 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Participants (%) with a vaginal and/or rectal detection of Group B Streptococcus. | 6 months
  Percentage of participants with a vaginal and/or rectal detection of Group B Streptococcus at the end of the study.

SECONDARY OUTCOMES:
Microbiota of vaginal exudates | 6 months
  Composition of the microbiota of vaginal exudates
Microbiota of rectal exudates | 6 months
  Composition of the microbiota of vaginal exudates
Premature membrane rupture | 7 months
  Percentage of participants with premature rupture of the membranes
Premature detachment of the placenta | 7 months
  Percentage of participants with premature delivery
Premature delivery | 7 months
  Percentage of participants with premature delivery
Pregnancy complications | 7 months
  Percentage of participants with pregnancy complications
Newborns with early onset sepsis | 7 months
  Percentage of newborns with early onset sepsis
Newborns with late onset sepsis | 7 months
  Percentage of newborns with late onset sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Susana Manzano, PhD, Study Chair — ProbiSearch SL
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Galvez A, Di Az de Teran E, Espinosa JA, Perez-Pedregosa J, Bartha-Rasero JL, Del Valle JG, Cuerva MJ, Jimenez E, Badiola C. Ligilactobacillus salivarius V4II-90 eradicates Group B Streptococcus colonisation during pregnancy: a randomised, double-blind, placebo-controlled trial. Benef Microbes. 2024 Jun 28;15(4):387-396. doi: 10.1163/18762891-bja00021. PMID 38955352